CLINICAL TRIAL: NCT00045721
Title: Phase I Trial of GLIADEL and O(6)-Benzylguanine in Pediatric Patients With Recurrent Malignant Gliomas
Brief Title: Carmustine Implants and O(6)-Benzylguanine in Treating Children With Recurrent Malignant Glioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James M. Boyett/PBTC Operations and Biostatistics Center Executive Director, Pediatric Brain Tumor Consortium
Purpose: Treatment
Other Study IDs: CDR0000257268; PBTC-009
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent childhood cerebral astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma | interventions — O(6)-benzylguanine; Carmustine; Chemotherapy, Adjuvant; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: O6-benzylguanine
Drug: polifeprosan 20 with carmustine implant
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemotherapy placed into the surrounding tissue after surgery to remove the tumor may kill any remaining tumor cells. O(6)-benzylguanine may increase the effectiveness of carmustine by making tumor cells more sensitive to the drug.

PURPOSE: Phase I trial to study the safety of combining O(6)-benzylguanine with carmustine implants in treating children who have recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose of O(6)-benzylguanine that reliably inhibits alkylguanine-DNA alkyltransferase activity in pediatric patients with recurrent malignant glioma.
* Describe the toxic effects of O(6)-benzylguanine with carmustine implant (Gliadel) in these patients.
* Investigate antitumor response in patients treated with this regimen.
* Characterize the pharmacokinetics of O(6)-benzylguanine when administered continuously over a 9-day period.

OUTLINE: This is a multicenter, dose-escalation study of O(6)-benzylguanine.

Patients receive O(6)-benzylguanine (O6-BG) IV over 1 hour immediately followed by O6-BG IV continuously for 9 days. Two days after initiation of continuous infusion of O6-BG, patients undergo maximal tumor debulking. At the time of surgery, patients receive up to 8 polifeprosan 20 wafers with carmustine (Gliadel) implanted into the resection cavity.

Cohorts of up to 14 patients receive escalating doses of continuous infusion O6-BG until the optimally biologically effective dose (BED) is determined. The BED is defined as the dose at which at least 11 of 14 patients meet the target of complete suppression of alkylguanine-DNA alkyltransferase levels.

Patients are followed at day 11, at weeks 2, 4, 6, 8, and 12, at months 6, 9, and 12, every 6 months for 4 years, and then annually for 5 years.

PROJECTED ACCRUAL: Approximately 20 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed progressive supratentorial anaplastic astrocytoma or glioblastoma multiforme
* No multifocal disease or leptomeningeal dissemination of tumor
* No evidence of tumor crossing midline
* Limited intraventricular involvement
* Measurable unilateral mass at least 10 mm by contrast-enhanced MRI
* Received prior involved-field radiotherapy as a component of prior therapy
* Amenable to and in need of significant debulking

PATIENT CHARACTERISTICS:

Age

* 3 to 21

Performance status

* Karnofsky 60-100% OR
* Lansky 60-100%

Life expectancy

* More than 8 weeks

Hematopoietic

* Absolute neutrophil count greater than 1,000/mm3*
* Platelet count greater than 100,000/mm3*
* Hemoglobin greater than 8 g/dL (transfusions allowed) NOTE: * Transfusion independent

Hepatic

* Bilirubin no greater than 1.5 times normal
* AST and ALT less than 3 times normal
* Albumin at least 2 g/dL
* No overt hepatic disease

Renal

* Creatinine clearance no greater than 1.5 times normal OR
* Glomerular filtration rate greater than 70 mL/min
* No overt renal disease

Cardiovascular

* No overt cardiac disease

Pulmonary

* No overt pulmonary disease

Other

* Neurological deficits must be stable for at least the past week
* No uncontrolled infection
* No known hypersensitivity to nitrosoureas or polyethylene glycol
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 6 months since prior bone marrow transplantation
* More than 2 weeks since prior colony-stimulating growth factors (e.g., filgrastim (G-CSF), sargramostim (GM-CSF), or epoetin alfa)

Chemotherapy

* No more than 2 prior cytotoxic chemotherapy regimens
* No more than 3 prior chemotherapy regimens total
* More than 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas) and recovered
* Prior systemic carmustine (or other nitrosourea) allowed provided patient did not experience non-hematopoietic grade III/IV toxicity

Endocrine therapy

* Concurrent dexamethasone allowed if on a stable dose for at least the past week

Radiotherapy

* See Disease Characteristics
* At least 3 months since prior radiotherapy
* No prior craniospinal irradiation for metastatic disease

Surgery

* See Disease Characteristics
* Prior biopsy or cytoreductive surgery allowed

Other

* Concurrent anticonvulsants allowed
* No other concurrent anticancer or investigational drugs

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2003-03; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Biologically effective dose of O(6)-benzylguanine administered continuously in pediatric patients with recurrent malignant glioma
Toxicities associated with the administration of O(6)-benzylguanine and carmustine implants.

SECONDARY OUTCOMES:
Tumor response

CONTACTS AND LOCATIONS:
Overall Officials: Ian F. Pollack, MD, Study Chair — University of Pittsburgh
Locations (9):
- United States (9):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer Center, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington